CLINICAL TRIAL: NCT02843698
Title: Effects of Dexmedetomidine on Oxygenation and Lung Mechanics in Morbidly Obese Patients Undergoing Bariatric Operations: A Randomized Controlled Trial
Brief Title: Effects of Dexmedetomidine on Oxygenation and Lung Mechanics in Morbidly Obese Patients Undergoing Bariatric Operations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-12-2016
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Restrictive Lung Disease
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will receive either, Dexmedetomidine (Precedex, Hospira, Lake forest, IL, USA) in a dose of (1ug/Kg LBW) bolus followed by 0.5ug/Kg continuous infusion for one hour
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients will receive normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion was previously reported to improve oxygenation and lung dynamics in patients with obstructive lung diseases. In our study we are going to investigate its effect on oxygenation and lung dynamics in restrictive lung disease
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Normal saline — Normal saline
  Other Names: Saline
  Arms: Control group

SUMMARY:
The study aims to investigate the effect of dexmedetomidine on oxygenation and lung mechanics in morbidly obese patients

DETAILED DESCRIPTION:
The patients of interest are morbid obese patients scheduled for bariatric surgery. Dexmeditomidine will be infused intraoperatively after induction of anesthesia. lung mechanics (dead space and compliance) as well as oxygenation (PF ratio) will be monitored intraoperatively and postoperatively

ELIGIBILITY:
Inclusion Criteria:

- Morbid obese (body mass index > 40) with documented restrictive lung disease scheduled to bariatric operation.

Exclusion Criteria:

* Heart failure
* ِِِِArrhythmia
* Heart block
* Severe liver or kidney impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 2 hours
  assessed by P/F ratio

SECONDARY OUTCOMES:
Lung mechanics | 2 hours
  lung compliance and dead space
arterial blood pressure | 2 hours
  arterial blood pressure measured in mmHg
plateau airway pressure | 2 hours
  plateau airway pressure measured in cmH2o
heart rate | 2 hours
  number of heart beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasanin A, Taha K, Abdelhamid B, Abougabal A, Elsayad M, Refaie A, Amin S, Wahba S, Omar H, Kamel MM, Abdelwahab Y, Amin SM. Evaluation of the effects of dexmedetomidine infusion on oxygenation and lung mechanics in morbidly obese patients with restrictive lung disease. BMC Anesthesiol. 2018 Aug 14;18(1):104. doi: 10.1186/s12871-018-0572-y. PMID 30103679